CLINICAL TRIAL: NCT05454657
Title: A Pilot Study of Ambulatory Heart Rate Variability Biofeedback for Substance Use Disorder
Brief Title: Heart Rate Variability Biofeedback for Substance Use Disorder: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Colorado State University (Other)
Responsible Party: Principal Investigator, David Eddie, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022P001496
Record Dates: First submitted 2022-07-04; First posted 2022-07-12 (Actual); Results first posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Substance Use Disorders
Keywords: Heart rate variability biofeedback; Just in time; Autonomic nervous system; Substance use disorder; Addiction recovery
MeSH Terms: conditions — Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Heart rate variability biofeedback + treatment as usual vs. treatment as usual only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Heart rate variability biofeedback + treatment as usual (Experimental): The experimental group participated in 8 weeks of Heart Rate Variability Biofeedback (HRVB) practice using the Lief HRVB Smart Patch and smartphone app + treatment as usual. Participants were asked to, 1) wear the Lief Smart Patch for at least 8 hours per day, 2) do 10mins of scheduled HRVB practice daily, and 3) do at least 5mins per day of HRVB practice in-the-moment when negative affect/craving arose, or in response to just-in-time prompts to do brief bursts of HRVB when the device sensed autonomic arousal indicative of stress.
  Interventions: Device: Heart rate variability biofeedback + treatment as usual; Behavioral: Treatment as usual only
- Treatment as usual only (Active Comparator): The control group participated in 8 weeks of treatment as usual only.
  Interventions: Behavioral: Treatment as usual only

INTERVENTIONS:
Device: Heart rate variability biofeedback + treatment as usual — Heart rate variability biofeedback is a biobehavioral intervention involving rhythmic breathing at resonance frequency (RF) that stimulates the baroreflex and increases heart rate variability.
  Arms: Heart rate variability biofeedback + treatment as usual
Behavioral: Treatment as usual only — Treatment as usual may include any outpatient substance use disorder treatment or mutual-help group participation.

SUMMARY:
Heart rate variability biofeedback (HRVB) is an biobehavioral intervention involving rhythmic breathing at resonance frequency that stimulates cardiovascular regulatory systems to help individuals better regulate affect and bolster cognitive control. This intervention has already shown its potential as a substance use disorder (SUD) treatment tool, but practical limitations of its accessibility, labor intensiveness, and cost have previously prevented this intervention from going to scale. Second-generation, ambulatory HRVB technology, however, has overcome these limitations and now allows patients to practice HRVB in-the-moment when its needed most. This study is testing the efficacy of second-generation, ambulatory HRVB for the first time with individuals with SUD.

DETAILED DESCRIPTION:
Alcohol and other drug use (AOD) lapses in early substance use disorder (SUD) recovery typically arise from interactions between aversive affective states and stressors that together elicit urges to use. A central goal of first-line cognitive-behavioral SUD treatments is to strengthen affective and cognitive control to increase individuals' ability to override impulses to use AOD. Yet certain automatic physiological processes compromised by SUD dynamically interact with internal affective states and environmental cues to undermine effortful cognitive control and outcompete cognitive goals to avoid substance use.

Heart rate variability biofeedback (HRVB) is a biobehavioral intervention involving rhythmic breathing at resonance frequency (RF) that stimulates the body's baroreflex mechanism to offset these psychophysiological deficits. The autonomic normalization effected by RF breathing is thought to bolster cognitive control efforts by interrupting or dampening automatic-visceral reactions that can undermine treatment gains, and in doing so support better decision-making, motivation, reductions in craving, and shifts in attention allocation.

Previous studies of HRVB have focused on positive behavioral effects that accrue over a series of weeks or months, rather than 'in-the-moment'. These chronic behavior changes, although clinically valuable, are labor and time intensive to elicit, reducing the likelihood of large-scale uptake of the intervention. Further, first-generation HRVB's regular daily practice model is likely to only partially mitigate the intense momentary bouts of emotion dysregulation that are triggers for AOD use in those in early SUD recovery. In contrast, recent studies have demonstrated that a brief exposure to RF breathing in anticipation of psychosocial stress, or during induced stress, helps to control physiological arousal, reduce state anxiety, and improve cognitive performance. It is posited that such bursts of in-the-moment HRVB practice could serve as a potent SUD treatment tool that helps individuals self-regulate emotions when needed most.

Recent advances in the field have given rise to small, lightweight, wearable biosensors that can allow wearers to do HRVB on-the-go. These devices also have the capacity to function as a just-in-time intervention by prompting in-the-moment HRVB practice when autonomic hyperarousal is detected, to buffer salient triggers and urges to use AOD. This research builds on a body of preliminary work speaking to HRVB's potential as an addendum to first-line SUD treatments by exploring for the first time in this disorder this second-generation, ambulatory, HRVB technology. Specific aims of this research include, 1) assessing ambulatory HRVB's uptake by individuals with SUD, 2) testing day-level effects of in-the-moment HRVB practice on affective states and substance use, and 3) testing the accumulative effects of scheduled daily HRVB practice, in-the-moment HRVB practice, and their combination, on substance use.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Own a smartphone
* English proficiency
* DSM 5 diagnosis of substance use disorder
* In the first year of a current substance use disorder recovery attempt with a goal of total alcohol and other drug abstinence

Exclusion Criteria:

* Medical history of severe cardiac arrhythmia
* Active psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2025-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Eddie, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eddie D, Nguyen M, Zeng K, Mei S, Emery N. Heart Rate Variability Biofeedback for Substance Use Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2025 Dec 1;82(12):1177-1185. doi: 10.1001/jamapsychiatry.2025.2700. PMID 41032322

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a phase II, randomized clinical trial involving 8 weeks of outpatient treatment. Enrollment occurred virtually in the US from January 4 2023 to June 2024. Of 238 potential participants assessed, 120 treatment-seeking participants with an SUD were randomized.
Pre-assignment Details: All enrolled participants were assigned to a group.
Groups:
- Heart Rate Variability Biofeedback + Treatment as Usual: The experimental group participated in 8 weeks of Heart Rate Variability Biofeedback practice using the Lief Heart Rate Variability Biofeedback Smart Patch and smartphone app + treatment as usual. Participants were asked to, 1) wear the Lief Smart Patch for at least 8 hours per day, 2) do 15mins of scheduled Heart Rate Variability Biofeedback practice daily, and 3) use it as needed in response to negative affect in-the-moment.
Period: Overall Study
Arm/Group | Heart Rate Variability Biofeedback + Treatment as Usual | Treatment as Usual Only
Started | 70 | 50
Completed | 65 | 50
Not Completed | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Heart Rate Variability Biofeedback + Treatment as Usual | Treatment as Usual Only | Total
Number analyzed (Participants) | 65 | 50 | 115
Age, Continuous [Mean (Standard Deviation); unit: Years] — Five experimental group participants were excluded from the baseline analyses; four failed to comply with the study protocol and one was found to be ineligible after study enrollment.
  Years | 46.18 (12.08) | 46.18 (11.04) | 46.18 (11.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 29 | 69
  Male | 25 | 21 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 4 | 11
  White | 51 | 44 | 95
  More than one race | 4 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 61 | 44 | 105
  Unknown or Not Reported | 0 | 0 | 0
Perceived Stress Scale [Mean (Standard Deviation); unit: Units on a scale] — Scale range = 0-25; higher scores indicate greater stress
  Units on a scale | 14.83 (2.97) | 14.20 (3.30) | 14.56 (3.12)
Patient-Reported Outcomes Measurement Information System (PROMIS) - Anxiety 6a [Mean (Standard Deviation); unit: Units on a scale] — Scale range = 6-30; higher scores indicate greater anxiety
  Units on a scale | 16.20 (5.76) | 16.35 (5.19) | 16.26 (5.50)
Patient-Reported Outcomes Measurement Information System (PROMIS) - Depression 6a [Mean (Standard Deviation); unit: Units on a scale] — Scale range = 6-30; higher scores indicate greater depression
  Units on a scale | 14.71 (6.48) | 13.72 (5.47) | 14.28 (6.06)

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate Variability Biofeedback Engagement
Description: Number of participants with ≥50% daily-practice adherence to the study practice target of 15 minutes per day, inclusive of scheduled and self-initiated HRVB practice
Time Frame: 8 weeks
Population: An additional three participants were excluded from the within-treatment EMA analyses because they completed <10% of surveys (final within treatment n=112; 64 experimental; 48 controls).
Measure: Count of Participants; unit: Participants
Arm/Group | Heart Rate Variability Biofeedback + Treatment as Usual | Treatment as Usual Only
Number analyzed (Participants) | 64 | 48
Participants | 15 | 0

2. Primary Outcome: Day-level Negative Affect
Description: Average day-level score reported; Range = 0-10; higher values denote greater negative affect
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Heart Rate Variability Biofeedback + Treatment as Usual | Treatment as Usual Only
Number analyzed (Participants) | 64 | 48
Scores on a scale | 2.96 (2.07) | 3.36 (2.13)
Statistical Analysis 1: Comparison: Heart Rate Variability Biofeedback + Treatment as Usual vs Treatment as Usual Only; To test the effect of HRVB vs control on negative affect, a multilevel model was estimated where study day predicted mean negative affect that same day (L1; within-person), while controlling for day-of-the-week. At Level 2 (between-person), treatment condition and sex were included as predictors of negative affect. The focal effects were the main effect of treatment condition (L2) and cross-level interactions between study day (L1) and treatment condition (L2) predicting daily negative affect; Test type: Superiority; p < .05, Mixed Models Analysis; Slope = -.01, 95% CI 2-sided [-.015 to -.008] — Cross-level interaction effect of Study Day X Treatment Group

3. Primary Outcome: Day-level Positive Affect
Description: Average day-level score reported; Range = 0-10; higher values denote greater positive affect
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Heart Rate Variability Biofeedback + Treatment as Usual | Treatment as Usual Only
Number analyzed (Participants) | 64 | 48
Scores on a scale | 5.26 (1.97) | 5.02 (1.92)
Statistical Analysis 1: Comparison: Heart Rate Variability Biofeedback + Treatment as Usual vs Treatment as Usual Only; To test the effect of HRVB vs. control on positive affect, a multilevel model was estimated where study day predicted mean positive affect that same day (L1; within-person), while controlling for day-of-the-week. At Level 2 (between-person), treatment condition and sex were included as predictors of positive affect. The focal effects were the main effect of treatment condition (L2) and cross-level interactions between study day (L1) and treatment condition (L2) predicting daily positive affect; Test type: Superiority; p < .05, Mixed Models Analysis; Slope = .01, 95% CI 2-sided [-.677 to .857] — Cross-level interaction effect of Study Day X Treatment Group

4. Primary Outcome: Day-level Craving
Description: Average day-level score reported; Range = 0-10; higher values denote greater craving
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Heart Rate Variability Biofeedback + Treatment as Usual | Treatment as Usual Only
Number analyzed (Participants) | 64 | 48
Scores on a scale | 2.32 (2.65) | 2.25 (2.77)
Statistical Analysis 1: Comparison: Heart Rate Variability Biofeedback + Treatment as Usual vs Treatment as Usual Only; To test the effect of HRVB vs. control on craving, a multilevel model was estimated where study day predicted mean craving that same day (L1; within-person), while controlling for day-of-the-week. At Level 2 (between-person), treatment condition and sex were included as predictors of craving. The focal effects were the main effect of treatment condition (L2) and cross-level interactions between study day (L1) and treatment condition (L2) predicting daily craving; Test type: Superiority; p < .05, Mixed Models Analysis; Slope = -.02, 95% CI 2-sided [-.026 to -.014] — Cross-level interaction effect of Study Day X Treatment Group

5. Primary Outcome: Day-level Substance Use
Description: Percent participants reporting any day-level substance use
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Heart Rate Variability Biofeedback + Treatment as Usual | Treatment as Usual Only
Number analyzed (Participants) | 64 | 48
Participants | 6 | 5
Statistical Analysis 1: Comparison: Heart Rate Variability Biofeedback + Treatment as Usual vs Treatment as Usual Only; To test the effect of HRVB vs. control on AOD use A Bayesian logistic multilevel model was estimated where study day predicted AOD use that same day (L1; within-person), while controlling for day-of-the-week. At Level 2 (between-person), treatment condition and sex were included as predictors of AOD use. The focal effects were the main effect of treatment condition (L2) and cross-level interactions between study day (L1) and treatment condition (L2) predicting daily AOD use; Test type: Superiority; p < 0.05, Mixed Models Analysis — 95% Bayesian Credible Intervals Intervals are used to determine significance, and significance is represented by credible intervals that do not include 0 or 1.00 when odds ratios are calculated; Odds Ratio (OR) = 0.36, 95% CI 2-sided [0.245 to 0.543] — Main effect of treatment group

6. Primary Outcome: 8-week Substance Use
Description: Mean percent days abstinent over the 8-week intervention period
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of days abstinent
Arm/Group | Heart Rate Variability Biofeedback + Treatment as Usual | Treatment as Usual Only
Number analyzed (Participants) | 64 | 48
percentage of days abstinent | 91.79 (18.03) | 90.33 (16.99)
Statistical Analysis 1: Comparison: Heart Rate Variability Biofeedback + Treatment as Usual vs Treatment as Usual Only; Two-sample t test with unequal variances; Test type: Equivalence — Two-sample t test with unequal variances; p = .660, t-test, 2 sided; Unequal variances were specified as part of the model; Mean Difference (Net) = -1.47, 95% CI 2-sided [-8.07 to 5.13], Standard Error of Mean 3.33

7. Primary Outcome: Odds Ratio of Within-day Association Between AOD Craving and AOD Use
Description: Within-day association between alcohol and other drug (AOD) craving earlier in the day and the odds of AOD use later that same day
Time Frame: 8 weeks
Population: To test the moderating effects of HRVB on the within-day associations between craving and AOD use, we estimated a Bayesian logistic multilevel model with an unstructured variance-covariance matrix where craving earlier in the day predicted AOD use later that same day (L1; lagged within-person). The focal effect of interest was a cross-level interaction between craving earlier in the day (L1) and treatment condition (L2) predicting AOD use later that same day.
Measure: Number; unit: Odds ratio
Arm/Group | Heart Rate Variability Biofeedback + Treatment as Usual | Treatment as Usual Only
Number analyzed (Participants) | 64 | 48
Odds ratio | 0.84 | 1.00

8. Secondary Outcome: Change Craving
Description: Change in craving measured by ecological momentary assessment over the 8-week intervention period, modeled using time-varying effects modeling (TVEM).
Time Frame: 8 weeks
Reporting Status: Not Posted, anticipated posting 2026-03

9. Secondary Outcome: Change Positive Affect
Description: Change in positive affect measured by ecological momentary assessment over the 8-week intervention period, modeled using time-varying effects modeling (TVEM).
Time Frame: 8 weeks
Reporting Status: Not Posted, anticipated posting 2026-03

10. Secondary Outcome: Change Negative Affect
Description: Change in negative affect measured by ecological momentary assessment over the 8-week intervention period, modeled using time-varying effects modeling (TVEM).
Time Frame: 8 weeks
Reporting Status: Not Posted, anticipated posting 2026-03

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Heart Rate Variability Biofeedback + Treatment as Usual | Treatment as Usual Only
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/50
Other Adverse Events (participants affected / at risk) | 0/70 | 0/50

LIMITATIONS AND CAVEATS:
Limitations include: (1) a modest sample size and no placebo group, reflecting the phase II stage of the trial; (2) focus on individuals in their first year of abstinence-based SUD recovery, enhancing relevance for this group but limiting generalizability; (3) lack of follow-up; and (4) testing only the hypothesized moderation effect of HRVB on the craving-AOD use relationship, without examining other mechanisms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-27): https://cdn.clinicaltrials.gov/large-docs/57/NCT05454657/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-29): https://cdn.clinicaltrials.gov/large-docs/57/NCT05454657/ICF_001.pdf